CLINICAL TRIAL: NCT03083678
Title: A Phase 2, Single Arm, European Multi-center Trial Evaluating the Efficacy of Afatinib As First-line or Later-line Treatment in Advanced Chordoma.
Brief Title: Afatinib in Locally Advanced and Metastatic Chordoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Chordoma Foundation (Other); Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, HansGelderblom, Prof. Dr., Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.277
Record Dates: First submitted 2017-02-10; First posted 2017-03-20 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Chordoma
Keywords: EGFR; Afatinib
MeSH Terms: conditions — Chordoma | interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Afatinib (Experimental): Afatinib active treatment.
  Interventions: Drug: Afatinib

INTERVENTIONS:
Drug: Afatinib — Afatinib will be given daily in a dose of 40 mg orally in a 4 week cycle until disease progression or patient withdrawal.
  Other Names: Giotrif

SUMMARY:
In this phase 2, single arm trial patients with locally advanced or metastatic, pathologically proven, EGFR expressing chordoma will be treated with afatinib. Two cohorts of patients will be included: 20 first line patients and 20 second or further line patients. The treatment will be given in 4 week cycles until disease progression. Median PFS according to RECIST 1.1 will be evaluated. The objective is to increase the median PFS ≥ 12 months in first-line treatment cohort and ≥ 9 months in later-line treatment cohort. Additional exploratory research will be performed, consisting of a pharmacokinetic study and translational studies on EGFR pathway activation and signalling on blood and tumor samples.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic, pathologically proven, EGFR expressing chordoma, not amenable for local therapies
* Patients of 18 years and up
* Documented radiographic progression of disease according to RECIST 1.1 criteria in last 6 months
* ECOG Performance status ≤ 2
* Adequate bone marrow function (Hb ≥ 6.0 mmol/L, absolute neutrophil count ≥ 1.5 x 109/L, platelets ≥ 75 x 109/L)
* An adequate renal function with GFR ≥ 45 ml/min calculated by Cockroft-Gault formula
* Total Bilirubin ≤ 1.5 times upper limit of normal (ULN) (Patients with Gilbert's syndrome total bilirubin must be ≤4 times institutional upper limit of normal).
* Aspartate amino transferase (AST) or alanine amino transferase (ALT) ≤ 3 times ULN (if related to liver metastases ≤ 5 times ULN)
* Ability to swallow medication
* Recovered from any previous therapy related toxicity to ≤ grade 1 at study entry (except for stable sensory neuropathy ≤ grade 2 and alopecia)
* Availability of archival tumor material for central review (if not please obtain a new tumor biopsy)
* Written signed informed consent
* Ability to adhere to the study visits and all protocol requirements

Exclusion Criteria:

* Life expectancy of less than 3 months
* No measurable lesions according to RECIST 1.1
* Known hypersensitivity to afatinib
* Major surgery less than 4 weeks prior to start of treatment
* Previous treatment with any other investigational agents within 14 days of first day of study drug dosing
* History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure NYHA classification of ≥ 3, unstable angina or poorly controlled arrhythmia as determined by the investigator. Myocardial infarction within 6 months prior to inclusion.
* Known pre-existing interstitial lung disease
* Any history or presence of poorly controlled gastrointestinal disorders that could affect the absorption of the study drug (e.g. Crohn's disease, ulcerative colitis, chronic diarrhea, malabsorption)
* Known active hepatitis B infection (defined as presence of HepB sAg and/ or Hep B DNA), active hepatitis C infection (defined as presence of Hep C RNA) and/or known HIV carrier.
* Systemic anti-cancer therapy within 28 days prior to the first dose of study drug , or radiotherapy to an index (or target)lesion within 21 days prior to the first dose of study drug
* Requiring treatment with any of the prohibited concomitant medications listed in Section 6.3.9 that cannot be stopped for the duration of trial participation
* Pregnant or lactating women
* Other invasive malignancies diagnosed within the last 5 years, except non-melanoma skin cancer and localized cured prostate and cervical cancer
* Any history of or concomitant condition that, in the opinion of the Investigator, would compromise the patient's ability to comply with the study or interfere with the evaluation of the efficacy and safety of the test drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Median PFS according to RECIST 1.1 criteria on afatinib treatment (first-line cohort) | From date of start treatment until date of first documented of progression or withdrawal (through study completion, an average of 1 year).
  The objective is to increase the median PFS ≥ 12 months in first-line treatment cohort.
Median PFS according to RECIST 1.1 criteria on afatinib treatment (second or later line cohort) | From date of start treatment until date of first documented of progression or withdrawal (through study completion, an average of 1 year).
  The objective is to increase the median PFS ≥ 9 months in later-line treatment cohort.
Quality of life assessment by EORTC QLC-30 questionnaire. | From date of start treatment until date of first documented of progression of withdrawal (through study completion, an average of 1 year).
  Change from baseline in EORTC QLC-30 questionnaire score.
Quality of life assessment by Brief pain inventory short form | From date of start treatment until date of first documented of progression of withdrawal (through study completion, an average of 1 year).
  Change from baseline on Brief pain inventory short form score.

SECONDARY OUTCOMES:
Growth modulation index. | From date of start treatment until date of first documented of progression (through study completion, an average of 1 year).
  Time to progression during afatinib treatment (TTP2) divided by time to progression before start of this treatment TTP1 (= growth modulation index)
Toxicity determined by CTCAE v 4.03 criteria | From date of start treatment until date of first documented of progression or withdrawal (through study completion, an average of 1 year).
  Toxicity determined by CTCAE v 4.03 criteria
Overall survival. | Survival follow-up after end of treatment every 3 months for up to 2 years followed by contact at 3 years.
  Overall survival from start of afatinib treatment

OTHER OUTCOMES:
Translational research - EGFR pathway analysis in tumor tissue | From date of inclusion until date of first documented of progression or withdrawal (through study completion, an average of 1 year)
  EGFR status by FISH / immunohistochemistry
Translational research - Genome sequence analysis of available tumor samples | From date of inclusion until date of first documented of progression or withdrawal (through study completion, an average of 1 year)
  Genetic mutations by DNA whole genome sequencing of fresh samples
Translational research - circulating tumor DNA | Analysis on blood samples to be taken at baseline, cycle 4 day 1, cycle 7 day 1 and at end of treatment (within 30 days after last dose of study drug).
  Circulating chordoma tumor DNA identification by WGS and PCR
Translational research - circulating exosomes | Analysis on blood samples to be taken at different time points on cycle 1 day 1, cycle 1 day 15, cycle 3 day 1 and cycle 5 day 1.
  Circulating exosomes identification by PCR
Pharmacokinetic research | Analysis on blood samples to be taken at different time points on cycle 1 day 1, cycle 1 day 15, cycle 3 day 1 and cycle 5 day 1.
  Area under the curve

CONTACTS AND LOCATIONS:
Overall Officials: AJ Gelderblom, Prof, Principal Investigator — Leiden University Medical Center
Locations (3):
- Istituto Nazionale dei Tumori: Fondazione IRCCS, Milan, Italy
- Leiden University Medical Center, Leiden, Netherlands
- University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided